CLINICAL TRIAL: NCT04684134
Title: High-Risk Factors in Patients With Colorectal Polyps a Prospective Case-Control Study
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-020
Record Dates: First submitted 2020-11-30; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: patients with colorectal polyps
- control group: patients without intestinal diseases

SUMMARY:
This prospective case-control study aimed to analyze and summarize the high-risk factors and susceptible genes of patients with colorectal polyps. According to these high-risk factors, the investigators developed and validated a prediction model for colorectal polyps to identify high-risk individuals, in order to provide clinical basis for the etiology research and the establishment of effective preventive measures.

DETAILED DESCRIPTION:
A large cohort of eligible participants were included in the analysis, and classified into derivation and validation cohorts at a ratio of 7:3. Demographic and clinicopathological characteristics of participants were utilized to develop a prediction model for colorectal polyps. In the derivation cohort, the LASSO regression method was applied to filter variables and select the most useful high-risk factors. Multivariate logistic regression analysis was used to identify potential predictors and then a prediction model was established. The predictive performance of the model was evaluated with respect to its discrimination, calibration and clinical usefulness.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥18 and ≤80 years old. Subject with complete data on demography and clinicopathology.

Exclusion Criteria:

- Subject with inflammatory bowel disease, enterophthisis, familial adenomatous polyposis, P-J syndrome and intestinal lymphoma.

A history of severe systemic diseases: liver cirrhosis, metabolic syndrome, chronic kidney disease, malignancy.

Subject taking blood lipid-lowering drugs, hormone or immunosuppressive agents. Unwillingness to cooperate with questionnaire survey. Lack of complete clinical data for analysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 2800 confirmed eligible participants, 18 to 80 years of age, including 2000 cases with colorectal polyps and 800 controls free of colorectal polyps, are enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Demographic and clinicopathological characteristics of participants with polyps | 1 year
  demographic and clinicopathological characteristics

SECONDARY OUTCOMES:
Independent high-risk factors of participants with polyps | 1 year
  high-risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oines M, Helsingen LM, Bretthauer M, Emilsson L. Epidemiology and risk factors of colorectal polyps. Best Pract Res Clin Gastroenterol. 2017 Aug;31(4):419-424. doi: 10.1016/j.bpg.2017.06.004. Epub 2017 Jun 28. PMID 28842051
- [Background] Bailie L, Loughrey MB, Coleman HG. Lifestyle Risk Factors for Serrated Colorectal Polyps: A Systematic Review and Meta-analysis. Gastroenterology. 2017 Jan;152(1):92-104. doi: 10.1053/j.gastro.2016.09.003. Epub 2016 Sep 14. PMID 27639804